CLINICAL TRIAL: NCT00497276
Title: A Prospective, Randomized Comparison of Ultrasound Versus Nerve Stimulation Guidance of Popliteal, Sciatic Catheter Placement After Major Foot and Ankle Surgery: Clinical Outcome and Cost Analysis
Brief Title: Comparison of Ultrasound and Nerve Stimulation Technique for Continuous Sciatic Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: National Board of Health, Denmark (Other Government)
Responsible Party: Danish Centre for Health Technology Assessment (DACEHTA), Danish Centre for Health Technology Assessment (DACEHTA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0-204-03-8/27
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Pain
Keywords: Adults; Anesthesia recovery period; Comparative study; Electric stimulation; Humans; Nerve blocks/methods/indications; Patient satisfaction; Peripheral nerves; Sciatic nerve/ultrasonography; Ultrasonography; Treatment outcome; Nerve blocks/economics
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Ultrasound guided placement of popliteal catheter
  Interventions: Procedure: placement of popliteal catheter
- II (Experimental): Nerve stimulation guided placement of popliteal catheter
  Interventions: Procedure: placement of popliteal catheter

INTERVENTIONS:
Procedure: placement of popliteal catheter — Bolus naropin 7,5 mg/ml 30 ml; infusion bupivacaine 2,5 mg/ml 5-10 ml/h

SUMMARY:
The most useful method to manage pain after major foot and ankle surgery is infusion of local anesthetic with a catheter close to the sciatic nerve in the popliteal space above the knee joint.

Inaccurate catheter placement and spread of local anesthetic account for most failures.

The most prevalent method to place the catheter is the traditional nerve stimulation technique relying on surface anatomic landmarks and electrical stimulation to localize the sciatic nerve. In recent years ultrasound technique has been applied to provide real-time, visual guidance of catheter placement.

The purpose of this randomized, controlled trial is to compare the success rate, patient acceptance and cost-effectiveness of the ultrasound and nerve stimulation techniques.

DETAILED DESCRIPTION:
Foot and ankle surgery is typically very painful for the first two days postoperatively due to surgical oedema. This pain is difficult to control with systemic analgesics. Pain relief with systemic analgesics requires high doses of intravenous opioids and is associated with breakthrough pain and adverse effects of opioids (sedation, nausea, vomiting, obstipation, urinary retention, mouth dryness, respiratory depression, pruritus, vertigo and visual disturbances).

Single-shot technique provides analgesia for two to 30 hours even using analgesics with prolonged effect (bupivacaine, levobupivacaine, ropivacaine). The duration of the block depends on the local analgesic and the anatomical location. Popliteal block with bupivacaine last up to 24 hours. Continuous, peripheral nerve block with catheter technique for two days minimizes the need for systemic analgesics and their adverse effects. Continuous, peripheral nerve block has gained popularity for foot and ankle surgery, because better analgesia is obtained compared to intravenous opioids, and similar analgesia with fewer adverse effects compared to epidural catheter technique.

Today the nerve stimulation technique is the most prevalent technique to introduce catheters for peripheral nerve blocks. The success rate for postoperative analgesia after foot and ankle surgery with popliteal catheters is variable - typically 70% in our department. The patients with catheter failure have severe postoperative pain, high opioid dosages, cognitive blurring, nausea, vomiting, reduced ambulation, increased surgical stress response and increased morbidity. Pain problems and adverse effects prolongs postoperative observation time and maybe also time to discharge.

Ultrasound technique was employed for peripheral nerve blocks for the first time in 1978. However the utility was technically limited. In recent years, the evolution of high-frequency transducers and mobile ultrasound units have facilitated the application of ultrasound-guided peripheral nerve blocks. This technique allows dynamic visualization of nerves, needle tip location and spread of local analgesic in real-time.

The empirical basis supporting the theoretical advantages of ultrasound-guided regional anesthesia consists mainly of observational studies. A few, randomized, controlled trials comparing ultrasound- and nerve stimulation technique favour the benefit of ultrasound concerning success rate, sensory onset time, duration of block, patient satisfaction and quality of block.

The purpose of this study is to establish whether ultrasound technique has higher success rate, better patient satisfaction and higher cost-effectiveness compared to electrical nerve stimulation using popliteal, sciatic catheters for postoperative analgesia after foot and ankle surgery.

ELIGIBILITY:
Inclusion Criteria:

elective posterior foot and/or ankle surgery

* calcaneus osteotomy
* subtalar arthrodesis
* total ankle arthroplasty
* ankle arthrodesis (non-arthroscopic) minimum age 18 years ASA I-III informed consent

Exclusion Criteria:

* coagulation disorders
* infection in the region of needle insertion
* systemic infection
* preoperative sciatic nerve neuropathy
* preoperative motor or sensory deficit in the operative extremity
* Charcot-Marie-Tooth disorder
* diabetic neuropathy
* severe peripheral vascular disease
* allergy to local anesthetics
* lack of understanding of the visual analogue scale
* communication problems
* dementia
* body mass index above 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Success rate: post-operative analgesia | First two post-operative days

SECONDARY OUTCOMES:
Time consumption of catheter placement | Before surgery
Duration of post-operative observation | After surgery
Pain score | First two post-operative days
Nausea score | First two post-operative days
Sensory block | First two post-operative days
Patient acceptance | First two postoperative days
Cost-effectiveness | Two days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Bendtsen, Ph.d., Principal Investigator — Department of Anesthesiology, Aarhus University Hospital, Norrebrogade, DK-8000 Aarhus C, Denmark
Locations (1):
- Department of Anesthesiology, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Ehlers L, Jensen JM, Bendtsen TF. Cost-effectiveness of ultrasound vs nerve stimulation guidance for continuous sciatic nerve block. Br J Anaesth. 2012 Nov;109(5):804-8. doi: 10.1093/bja/aes259. Epub 2012 Jul 31. PMID 22855632
- [Derived] Bendtsen TF, Nielsen TD, Rohde CV, Kibak K, Linde F. Ultrasound guidance improves a continuous popliteal sciatic nerve block when compared with nerve stimulation. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):181-4. doi: 10.1097/aap.0b013e31820d421f. PMID 21425514